CLINICAL TRIAL: NCT06110572
Title: (TESSERACT): Phase I/II Trial in ES-SCLC to Enhance Response to Atezolizumab Plus Chemotherapy With Total Body Irradiation (TBI)
Brief Title: Phase I/II Trial in ES-SCLC to Enhance Response to Atezolizumab Plus Chemotherapy With Total Body Irradiation
Acronym: TESSERACT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Evan Osmundson, MD, PhD, Associate Professor of Radiation Oncology, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICCTHOP2206; NCI-2023-08550 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma; Stage IV Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; atezolizumab; Etoposide; Whole-Body Irradiation; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (carboplatin, atezolizumab, etoposide, TBI, H-RT) (Experimental): Description INDUCTION PHASE: Patients receive carboplatin IV and atezolizumab IV on day 1 of each cycle and etoposide IV on days 1-3 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive TBI BID on day 18 or 19 of cycle 1 and beginning 2-3 days later, H-RT daily over 7 days in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Patients receive atezolizumab IV on day 1 of each cycle. Treatment repeats every 21 days for 12 cycles in the absence of disease progression or unacceptable toxicity.
  Patients also undergo CT and MRI throughout the trial.
  Interventions: Drug: Carboplatin; Biological: Atezolizumab; Drug: Etoposide; Radiation: Total Body Irradiation; Radiation: Hypofractionated Radiation Therapy; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Carboplatin — Given by IV
Biological: Atezolizumab — Given by IV
Drug: Etoposide — Given by IV
Radiation: Total Body Irradiation — Undergo Total Body Irradiation
Radiation: Hypofractionated Radiation Therapy — Undergo Hypofractionated Radiation Therapy
Procedure: Magnetic Resonance Imaging — Undergo Magnetic Resonance Imaging

SUMMARY:
This phase I/II trial studies the side effects, safety, and effectiveness of low dose radiation to the entire body (total body irradiation [TBI]) and higher dose radiation to known areas of cancer (hypofractionated radiation therapy [H-RT]) combined with atezolizumab and chemotherapy (carboplatin & etoposide) in treating patients with small cell lung cancer that has spread to disease sites outside of the lung (extensive stage). Extensive stage disease has historically been treated with chemotherapy alone with consideration of chest (thoracic) radiation therapy for those with response to chemotherapy, as well as consideration of preventative radiation therapy to the head (prophylactic cranial irradiation). Emerging evidence supports the synergistic interactions between immunotherapy and radiation therapy. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of tumor cells. Etoposide is in a class of medications known as podophyllotoxin derivatives. It blocks a certain enzyme needed for cell division and DNA repair and may kill tumor cells. Combining TBI and H-RT with atezolizumab and chemotherapy may improve response to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety of the addition of total body irradiation (TBI) and hypo-fractionated radiation (H-RT) to atezolizumab and chemotherapy in patients with extensive stage-small cell lung carcinoma (ES-SCLC).

II. Evaluate the efficacy of the addition of TBI and H-RT to atezolizumab and chemotherapy in patients with ES-SCLC.

SECONDARY OBJECTIVE:

I. Evaluate the progression free survival benefit and local and systemic control benefits of the addition of TBI and H-RT to atezolizumab and chemotherapy in patients with ES-SCLC.

OUTLINE:

INDUCTION PHASE: Patients receive carboplatin intravenously (IV) and atezolizumab IV on day 1 of each cycle and etoposide IV on days 1-3 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive TBI twice daily (BID) on day 18 or 19 of cycle 1 and beginning 2-3 days later, H-RT daily over 7 days in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Patients receive atezolizumab IV on day 1 of each cycle. Treatment repeats every 21 days for 12 cycles in the absence of disease progression or unacceptable toxicity.

Patients also undergo computed tomography (CT) and magnetic resonance imaging (MRI) throughout the trial.

After completion of study treatment, patients are followed up within 30 days and then every 3-4 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of informed consent
* Histologically documented or cytologically confirmed diagnosis of extensive stage small-celllung cancer with evaluable disease per RECIST v1.1 criteria. Patients may be considered extensive-stage based on M1 disease per AJCC 8th edition, OR may be clinically staged as extensive-stage disease based on anatomical extent that would preclude the use of standard radiotherapy fields as assessed by the treating radiation oncologist.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Lymphocyte count ≥ 0.5 x 10^9/L
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN, alanine aminotransferase (ALT) ≤ 2.5 x ULN and alkaline phosphatase ≤ 2.5 x ULN
* Creatinine ≤ 1.5 x ULN or calculated creatinine clearance (CrCl) ≥ 50 mL/min if creatinine (Cr) > 1.5 x ULN. GFR can also be utilized. If no local calculation guidance on CrCl, should be calculated according to Cockcroft-Gault Method
* International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless participant is receiving anticoagulation therapy. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen.
* Negative HIV test at screening, with the following exception: patients with positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200, and have an undetectable viral load
* Negative Hepatitis B surface antigen at screening
* Presence of brain metastases allowed (should undergo management with surgery and/or radiation therapy if symptomatic prior to TESSERACT radiation regimen; upfront cranial irradiation not mandatory on protocol if asymptomatic)
* Contraceptive use should be initiated or continued per guidance in labeling for approved chemotherapies
* Female patients must be non-pregnant and not breastfeeding
* Women of childbearing potential (WOCBP) must remain abstinent or use contraceptive methods with a failure rate of <1% per year during the treatment period and for 5 months after the final dose of atezolizumab. A woman is considered to be of childbearing potential if she is post-menarchal, has not reached a post-menopausal state (12 months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.

  * Examples of contraceptive methods with a failure rate of <1% per year include, bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptomthermal or postovulation methods) and withdrawal are not adequate methods of contraception.
  * With a female partner of childbearing potential who is not pregnant, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 5 months after the final dose of atezolizumab. Men must refrain from donating sperm during this same period.
  * With a pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 5 months after the final dose of atezolizumab to avoid exposing the embryo.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal.
* Eligible for immunotherapy-based systemic regimens per judgment of patient's study physician
* Able to submit written informed consent

Exclusion Criteria:

* Major surgery (requiring general anesthesia or at discretion of study physician) within 4 weeks prior to study enrollment that would prevent treatment with TESSERACT regimen
* Known clinically significant (per study physician) acute or chronic infections including HIV (per inclusion criteria above), hepatitis B virus (HBV), hepatitis C virus (HCV) or active tuberculosis (testing not required for tuberculosis [TB]). Patients with HCV must be on stable dose of antiviral therapy on study entry. Current treatment with antivirals for HBV is not allowed on study
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Uncontrolled hypertension (average systolic blood pressure greater than or equal to 140 or average diastolic blood pressure greater than or equal to 90 despite optimal medical therapy). Patients with hypertension (systolic blood pressure [SBP] ≥ 140 and/or diastolic blood pressure [DBP] ≥ 90) may enroll provided that an effective anti- hypertensive regimen is initiated.
* History of prior malignancy within 3 years of enrollment, except for adequately treated basal or squamous cell carcinoma of the skin, adequately treated carcinoma in situ (e.g. cervix or non- invasive bladder cancer) or other malignancy with minimal risk of metastasis or death (survival > 90% at 5 years)
* Receipt of prior courses of cytotoxic chemotherapy or anti-neoplastic biologic/immunotherapy for current malignancy (other than the current course of therapy). Patients may have undergone 1 cycle of 1st line of systemic therapy for SCLC prior to enrollment as long as the systemic therapy is congruent with what is included in the protocol and part of the current course of therapy.
* Prior radiotherapy that would preclude delivery of protocol- based radiotherapy to normal organ tolerance per patient's study physician
* Receipt of live attenuated vaccine within 28 days of cycle 1, day 1 (C1D1), and for 5 months after the last dose of atezolizumab.
* Use of prohibited concomitant drug
* Concurrent enrollment in another clinical trial (unless observational or within follow-up period)
* Known, pathologically confirmed malignant pleural effusions (diagnostic evaluation of pleural effusions are recommended but not required for study entry, especially if sampling is deemed technically challenging at discretion of treating physician)
* Uncontrolled pleural or pericardial effusion or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX) are allowed
* History of leptomeningeal disease
* Uncontrolled tumor-related pain: Patients requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy can undergo treatment with palliative radiotherapy prior to enrollment at discretion of treating physicians. Patients should be recovered from effects of radiation and there is no required minimum recovery period. Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) can be considered for loco-regional therapy at discretion of treating physician prior to enrollment.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, Inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid- replacement hormone are eligible for the study
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all the following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical steroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti- CTLA-4, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents including, but not limited to, interferon and interleukin 2 (IL-2) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents, within 2 weeks prior to initiation of study treatment with following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy are eligible for the study after Principal Investigator confirmation has been confirmed)
  * Patients who are receiving mineral corticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal sufficiency are eligible for the study.
  * Systemic steroids required during therapy for adverse event (AE) management are allowed.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months of the last dose of Atezolizumab. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Rates of treatment-related adverse events | Up to 30 days after completion of study treatment
  Graded by Common Terminology Criteria in Adverse Events version 5.0 (Grade 2-5).
Progression-free survival | From consent to the date of the first documentation of objective progressive disease (PD) or death due to any cause in the absence of documented PD, whichever occurs first, assessed up to 6 months
  Will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Kaplan-Meier estimates and associated statistics and corresponding 95% confidence intervals will be presented by treatment group

SECONDARY OUTCOMES:
Overall Survival | Up to 3 years
Overall Response Rate | Up to 3 years
  Defined according to RECIST/Immune-Modified (i)RECIST criteria.
Disease Control Rate | Up o 3 years
  Defined as the percentage of patients who have achieved complete response (CR), partial response (PR) or stable disease (SD). Exact Binomial test and 95% confidence interval (CI) will be used to assess DCR.
Intracranial Control Rate | Up to 3 years
  Defined as the percentage of patients who have SD, PR, CR or no evidence of disease (NED) in the brain. Exact Binomial test and 95% CI will be used to assess intracranial control rate.
Thoracic Control Rate | Up to 3 years
  Defined as the percentage of patients who have SD, PR, CR or NED in the thorax. Exact Binomial test and 95% CI will be used to assess thoracic control rate.
Duration of Response | Up to 3 years
  Defined as the length of time that patient continues to respond to treatment without progression according to RECIST 1.1/Immune-Related (ir)RECIST. 95% confidence interval will be constructed using Brookmeyer and Crowley method to assess DOR compared to historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Osmundson, MD, PhD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT06110572/ICF_000.pdf